CLINICAL TRIAL: NCT03160716
Title: A Multicenter, Open-Label, Prospective Study of Cannula Injection of Restylane Lyft With Lidocaine for Cheek Augmentation and the Correction of Age Related Midface Contour Deficiencies
Brief Title: Injection Technique Assessment of Restylane Lyft With Lidocaine for Cheek Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43USC1633
Record Dates: First submitted 2017-05-14; First posted 2017-05-19 (Actual); Results first posted 2019-05-15 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-05

CONDITIONS: Cheek Augmentation; Midface Contour Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Other)
  Interventions: Device: Restylane Lyft with Lidocaine

INTERVENTIONS:
Device: Restylane Lyft with Lidocaine — a sterile gel of hyaluronic acid (HA)

SUMMARY:
This is a multi-center, open-label, single-arm study to evaluate an injection tool with Restylane Lyft with Lidocaine for cheek augmentation and correction of age related midface contour deficiencies.

ELIGIBILITY:
Primary Inclusion Criteria:

* Subjects willing to comply with the requirements of the study and providing a signed written informed consent.
* Males or non-pregnant, non-breastfeeding females, 22 years of age or older.
* Mild to Substantial Midface Volume Loss

Primary Exclusion Criteria:

* Allergy or hypersensitivity to any injectable hyaluronic acid gel or to gram positive bacterial proteins
* Allergy or hypersensitivity to lidocaine or other amide-type anaesthetics, or topical anaesthetics or nerve blocking agents
* Undergone prior surgery to midface

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Facial Plastic and Cosmetic Surgery, Beverly Hills, California
  - Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California
  - Hessler Plastic Surgery, Palo Alto, California
  - Union Square Laser Dermatology, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones DH, Hessler J, Chapas A, Jonas B, Crider J, Chopra R. Microcannula Injection of Large Gel Particle Hyaluronic Acid for Cheek Augmentation and the Correction of Age-Related Midface Contour Deficiencies. Dermatol Surg. 2020 Apr;46(4):465-472. doi: 10.1097/DSS.0000000000002105. PMID 31490308

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 60
Completed | 59
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0
  Black/African American | 8
  Native Hawaiian/Other Pacific Islander | 1
  Asian | 6
  White | 43
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events [Safety]
Description: To assess the adverse events (incidence, intensity, and duration) of Restylane® Lyft with Lidocaine in conjunction with the use of a cannula.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 60
Participants | 5

2. Secondary Outcome: Number of Participants With Aesthetic Improvement
Description: To assess effectiveness using the Global Aesthetic Improvement Scale (GAIS). Responders defined as "Improved" or better on the GAIS as assessed by the investigator and participant at 2 weeks after week 16 re-treatment (visit only required for participants who received re-treatment at week 16).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 43
Participants | 43

3. Secondary Outcome: Number of Participants That Responded to Treatment
Description: To assess effectiveness using the 4-point Midface Volume Scale. Responder defined as at least a one point improvement from the baseline score at 2 weeks after week 16 re-treatment (visit only required for participants who received re-treatment at week 16).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 43
Participants | 43

4. Secondary Outcome: Subject Satisfaction
Description: To assess subject satisfaction with the treatment using the FACE-Q. Score range 1-100. The higher total score indicate greater subject satisfaction.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 59
score on a scale | 77.3 (23.5)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 5/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=60)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03160716/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03160716/SAP_001.pdf